CLINICAL TRIAL: NCT05982951
Title: A Comparative Study Between Ultrasound-guided Shoulder Block and Pericapsular Nerve Group Bock for Shoulder Arthroscopic Surgeries.
Brief Title: A Comparative Study Between Ultrasound Guided Shoulder Block and Pericapsular Nerve Group Bock for Shoulder Arthroscopic Surgeries: Double Blinded Randomized Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Kareem Mikhamer, Fellow lecturer of Anaesthesia, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GeneralCTHI
Record Dates: First submitted 2023-07-28; First posted 2023-08-09 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Efficacy of PENG Block Managing Perioperative Pain With Shoulder Arthroscopy Surgeries; Efficacy of Shoulder Block in Managing Perioperative Pain With Shoulder Arthroscopy Surgeries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The block will be performed by one investigator who is not participating in either data collection or analysis. Also the patient will be blinded .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder PENG block group (Active Comparator): Ultrasound-guided peri-capsular nerve block of the shoulder with 20ml of 0.25% bupivacaine between the supraspinatus muscle and deltoid muscle.
  Interventions: Procedure: Shoulder PENG block
- Shoulder block (Active Comparator): ultrasound guided axillary nerve block and suprascapular nerve block posterior approach with 10 ml 0.25% bupivacaine (total 20ml)
  Interventions: Procedure: Shoulder PENG block

INTERVENTIONS:
Procedure: Shoulder PENG block — Ultrasound guided insertion of a needle between subscapularis tendon and deltoid with injection of 10 mi 0.25% bupivacaine after confirming right plane of injection
  Other Names: Shoulder Block

SUMMARY:
Shoulder arthroscopic surgeries are one of the most common procedures performed daily in our practice. The arthroscopic techniques offer a less invasive option as Open repair does not offer a significantly better 2-year result in terms of stability, and furthermore, can negatively affect the recovery of the full range of motion of the shoulder. Open techniques Shoulder procedures are performed arthroscopically nowadays with fewer complications compared with open surgery.

Indications of shoulder arthroscopy are expanding and include biceps tears, labral tears, rotator muscle tears, subacromial impingements chondral injuries, loose bodies, early degenerative changes, adhesive capsulitis, shoulder instability and acromioclavicular osteoarthritis.

There are many regional anesthetic techniques used to control perioperative pain during arthroscopic procedures. Interscalene block results in effective shoulder surgery analgesia, but it is associated with various complications such as diaphragmatic paralysis due to the high incidence of phrenic nerve block.

The suprascapular nerve block combined with the axillary nerve block is non-inferior to conventional inter-scalene block except for the early recovery period with the advantage of lower incidence of dyspnea and discomfort.

. In a cadaveric anatomical study that the posterosuperior quadrant and the posteroinferior quadrant of the GHJ were innervated by the suprascapular nerve and the axillary nerve respectively. While the anterosuperior quadrant portion of the joint is sensory supplied by the subscapularis superior branch and the anteroinferior by the main branch of the axillary nerve. These anatomical data the possibility of a new block targeting the GHJ sensory branches. It was suggested that deep pericapsular infiltration of local anesthetic towards the subscapularis may cover the axillary and subscapularis branches that feed the anteroinferior and superior quadrants of the GHJ.

Recently, the pericapsular nerve group block of the shoulder joint as described in a case series including two cases underwent a humeral neck fracture fixation and Bankart arthroscopic repair with promising anesthesia and analgesia in selected shoulder surgeries.

DETAILED DESCRIPTION:
anesthetics Bleeding disorders receiving antiplatelet or anticoagulant drugs local infection at the site of local injection Intra articular infections

Sample size and methodology:

We will enroll 42 patients undergoing elective shoulder arthroscopy. They will be randomized and allocated into two groups; Group A and Group B. Group A will receive an ultrasound-guided PENG block and Group B will receive a shoulder block Sample size justification The sample size was calculated using Power Analysis and Sample Size software program (PASS) version 11.0.4 for Windows (2011) with time to first analgesic request as the primary outcome. Using the results published by Pani et al 2019 (8) with the mean time to first analgesic request in the shoulder block group was (5.9 ± 1.2 hours) Using a two-sided two-sample unequal-variance t-test, a sample size of 42 patients is needed to achieve 95% power to detect 20 % difference in time to a first analgesic request by using a two-sided hypothesis test with a significance level of 0.05.

Anticipated Results The application of pericapsular nerve group block in patients undergoing elective shoulder arthroscopic surgeries may improve the management of their perioperative pain.

Randomization:

The study subjects will be randomized by using block randomization using sealed concealed envelopes into two groups.

Data collection:

The patients will be observed for 24 hours postoperatively by a blinded investigator for the given block. All patients will receive one gram of acetaminophen intravenously every 8 hours as a part of the multimodal analgesia protocol.

The primary outcome will be the duration of analgesia (time to first rescue analgesia after administration of the block). Postoperative pain will be assessed using a 100 mm vertical visual analog score (VAS). The pain score will be recorded at 0, 1, 4, 8, 12, and 24 hours at rest (VASr) and movement (VASm). Morphine will be given intravenously if VASr, VASm, or both exceed 30mm in one milligram allequate with 5 minutes intervals till VAS is less than 30 mm or exceeds the safety dose of 30 mg in 4 hours.

Secondary outcomes:

Total fentanyl consumption as a rescue analgesia intraoperatively. Total morphine consumption in 24 hours postoperatively. Intraoperative hemodynamics mean arterial pressure and mean heart rate. length of stay in hospital Ability to perform physical rehabilitation program in the first 24 hours postoperatively.

postoperative sedation score using the Ramsey score patient satisfaction will be assessed by numerical score (1= very dissatisfied, 2= dissatisfied, 3=neither satisfied or dissatisfied, 4= satisfied, 5=very satisfied) postoperative nausea and vomiting (PONV) will be assessed using a 4 points numerical score (0=no PONV, 1= mild nausea, 2= severe nausea or vomiting once, 3= vomiting more than once)

Endpoint:

The observation of patients will be finished 24 hours postoperatively.

Results:

It will be recorded and analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II
* Age between 18 - 60
* unilateral elective shoulder arthroscopic surgery

Exclusion Criteria:

* Patient refusal
* Altered mental status or un-cooperative patients
* Hypersensitivity to local anesthetics
* Bleeding disorders
* receiving antiplatelet or anticoagulant drugs
* local infection at the site of local injection
* Intra articular infections

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-05 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia (time to first rescue analgesia) minutes | 24 hours after surgery
  Postoperative pain will be assessed using 100 millimeter vertical visual analog score (VAS) where (1-3) no pain, >3- 6) mild pain, and (>6 severe pain). The pain score will be recorded at 0, 1, 4, 8, 12, and 24 hours at rest (VASr) and movement (VASm). Morphine will be given intravenously if VASr, VASm, or both exceed 30mm in one milligram adequate with 5 minutes intervals till VAS be less than 30 mm or exceeds the safety dose of 30 mg in 4 hours.

SECONDARY OUTCOMES:
Total morphine consumption milligrams | 24 hours after surgery
  Total morphine consumption in 24 hours postoperatively.
Total fentanyl consumptions microgram | Intraoperative period
  Total fentanyl consumptions as a rescue analgesia intaoperatively
intraoperative hemodynamics | Intraoperative period
  Mean arterial blood pressure millimeter mercury , mean heart rate beat per minute
length of stay in hospital hours | 24 hours postoperative
  length of stay in hospital after surgery by hours
postoperative sedation | Immediate postoperative period
  Ramsey sedation Score
patient satisfaction | 24 hours postoperative
  numerical score (1= very dissatisfied, 2= dissatisfied, 3=neither satisfied or dissatisfied, 4= satisfied, 5=very satisfied)
postoperative nausea and vomiting (PONV) | 24 hours postoperative
  four points numerical score (0=no PONV, 1= mild nausea , 2= severe nausea or vomiting once, 3= vomiting more than once)

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher Teaching Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rockwood CA Jr. Shoulder arthroscopy. J Bone Joint Surg Am. 1988 Jun;70(5):639-40. No abstract available. PMID 3392055
- [Background] Severud EL, Ruotolo C, Abbott DD, Nottage WM. All-arthroscopic versus mini-open rotator cuff repair: A long-term retrospective outcome comparison. Arthroscopy. 2003 Mar;19(3):234-8. doi: 10.1053/jars.2003.50036. PMID 12627146
- [Background] Farmer KW, Wright TW. Shoulder arthroscopy: the basics. J Hand Surg Am. 2015 Apr;40(4):817-21. doi: 10.1016/j.jhsa.2015.01.002. Epub 2015 Feb 26. PMID 25726045
- [Background] Tran DQ, Elgueta MF, Aliste J, Finlayson RJ. Diaphragm-Sparing Nerve Blocks for Shoulder Surgery. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):32-38. doi: 10.1097/AAP.0000000000000529. PMID 27941477
- [Background] Neuts A, Stessel B, Wouters PF, Dierickx C, Cools W, Ory JP, Dubois J, Jamaer L, Arijs I, Schoorens D. Selective Suprascapular and Axillary Nerve Block Versus Interscalene Plexus Block for Pain Control After Arthroscopic Shoulder Surgery: A Noninferiority Randomized Parallel-Controlled Clinical Trial. Reg Anesth Pain Med. 2018 Oct;43(7):738-744. doi: 10.1097/AAP.0000000000000777. PMID 29659438
- [Background] Tran J, Peng PWH, Agur AMR. Anatomical study of the innervation of glenohumeral and acromioclavicular joint capsules: implications for image-guided intervention. Reg Anesth Pain Med. 2019 Jan 11:rapm-2018-100152. doi: 10.1136/rapm-2018-100152. Online ahead of print. PMID 30635516
- [Background] Kupeli I, Yazici Kara M. Anesthesia or analgesia? New block for shoulder surgery: pericapsular nerve group block. Braz J Anesthesiol. 2022 Sep-Oct;72(5):669-672. doi: 10.1016/j.bjane.2021.05.009. Epub 2021 Jun 9. PMID 34118263
- [Background] Pani N, Routray SS, Pani S, Mallik S, Pattnaik S, Pradhan A. Post-operative analgesia for shoulder arthroscopic surgeries: A comparison between inter-scalene block and shoulder block. Indian J Anaesth. 2019 May;63(5):382-387. doi: 10.4103/ija.IJA_65_19. PMID 31142882
- [Result] Grosh T, Elkassabany NM. Enhanced Recovery After Shoulder Arthroplasty. Anesthesiol Clin. 2018 Sep;36(3):417-430. doi: 10.1016/j.anclin.2018.04.006. PMID 30092938